CLINICAL TRIAL: NCT06700603
Title: Phase II Clinical Study of Irinotecan Liposome Combined with 5-FU/LV for the Patients with Advanced Pancreatic Cancer Who Failed to Receive Irinotecan-containing Regimens
Brief Title: Second-line Irinotecan Liposome Combination Regimen for Irinotecan-treated Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rui-hua Xu, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Rui-hua Xu, MD, PhD, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-PAAD-GD01
Record Dates: First submitted 2024-11-06; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
Keywords: Irinotecan; pancreatic; Irinotecan liposome
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Intervention Model Description: Cohort 1: Patients with imaging-confirmed progression during or within 3 months of completion of irinotecan treatment Cohort 2: Patients with imaging-proven disease progression 3 months after completion of irinotecan treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients with progression within 3 months of completion of irinotecan treament (Other): Cohort 1 was for patients who progressed within 6 months of the end of adjuvant therapy for early pancreatic cancer with a prior irinotecan regimen or for patients with advanced disease who had imaging-confirmed progression within 3 months of the end of first-line therapy.
  Interventions: Drug: Irinotecan liposome (Nal-IRI) in combination with 5-FU/sodium levofolinate
- Cohort 2: Patients with disease progression after 3 months of the end of irinotecan treatment (Other): Cohort 2 is for patients who have progressed more than 6 months after the end of adjuvant therapy for early pancreatic cancer on prior irinotecan regimens or more than 3 months after the end of first-line therapy for patients with advanced disease
  Interventions: Drug: Irinotecan liposome (Nal-IRI) in combination with 5-FU/sodium levofolinate

INTERVENTIONS:
Drug: Irinotecan liposome (Nal-IRI) in combination with 5-FU/sodium levofolinate — Irinotecan liposome (Nal-IRI) in combination with 5-FU/sodium levofolinate，Every 2 weeks until disease progression or patient develops intolerable toxicity

SUMMARY:
This study is a prospective, single-arm, two-cohort phase II clinical study. It is expected to enroll 48 patients with advanced or metastatic pancreatic cancer who have failed prior treatment with irinotecan-containing regimens, including two cohorts: cohort 1 for patients who have progressed within 6 months of the end of adjuvant therapy for early pancreatic cancer with a prior irinotecan regimen or for patients with imaging-confirmed progression within 3 months of the end of first-line therapy for advanced patients, and cohort 2 for patients who have progressed after more than Cohort 2 was for patients who had progressed more than 6 months after adjuvant treatment with previous irinotecan regimen for early-stage pancreatic cancer or more than 3 months after the end of first-line treatment for advanced-stage patients. The study was conducted at the Cancer Prevention and Control Center of Sun Yat-sen University. The study consists of a screening period (within 28 days), a treatment period (until disease progression or intolerable toxicity occurs in patients), and a follow-up period (12 months, safety follow-up and PFS follow-up). Subjects signed informed consent and underwent baseline examinations during the screening period, and patients who met the inclusion exclusion criteria entered the treatment period, and all subjects perfected the relevant examinations specified in the protocol during the treatment to observe safety, tolerability and efficacy. The same subject received only one dosing schedule during the study period. After the treatment period was completed, a follow-up period was entered.

DETAILED DESCRIPTION:
Evaluation of the efficacy and safety of irinotecan liposomes in combination with 5-FU/levulinic acid sodium in the treatment of patients with irinotecan-containing regimens for treated advanced pancreatic cancer Prospective, single-arm, dual-cohort phase II clinical study. Cohort 1: Patients with imaging-confirmed progression during or within 3 months of completion of irinotecan treatment Cohort 2: Patients with imaging-confirmed disease progression 3 months after completion of irinotecan treatment

ELIGIBILITY:
Inclusion Criteria:

* 1. patients are fully aware of the study, participate voluntarily and sign an informed consent form (ICF);
* 2. aged ≥18 years and ≤75 years;
* 3. histologically or cytologically confirmed as pancreatic ductal adenocarcinoma;
* 4. patients with advanced or metastatic pancreatic adenocarcinoma who have failed prior irinotecan-containing regimens and have no more than 3 prior lines of therapy.
* 5. patients with at least one measurable target lesion according to RECIST 1.1 criteria;
* 6. Eastern Cooperative Oncology Group (ECOG) physical status score: 0-1;
* 7. expected survival time ≥ 3 months;
* 8. absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 90 x 10^9/L and hemoglobin ≥ 90 g/L (not transfused with blood, blood products, or corrected with granulocyte colony-stimulating factor or other hematopoietic-stimulating factor in the 14 days prior to the laboratory test);
* 9. Liver and kidney function: serum creatinine ≤1.5 times the upper limit of normal; AST and ALT ≤2.5 times the upper limit of normal (≤5 times the upper limit of normal for patients with hepatic invasion); total bilirubin ≤1.5 times the upper limit of normal (≤3 times the upper limit of normal for patients with hepatic invasion);
* 10. Women of childbearing potential must have had a negative pregnancy test (serum) within 7 days prior to enrollment and be willing to use an appropriate method of contraception for the duration of the trial and for 6 months after the last administration of the test drug.

Exclusion Criteria:

* 1. hypersensitivity to any investigational drug or its components;
* 2. concomitant serious uncontrolled concurrent infections or other serious uncontrolled concomitant diseases, moderate or severe renal impairment; (e.g., progressive infections, uncontrollable hypertension, diabetes mellitus, etc.)
* 3. cardiac function and disease consistent with one of the following conditions

  1. Long QTc syndrome or QTc interval > 480 ms;
  2. Complete left bundle branch block, degree II or degree III atrioventricular block;
  3. Severe, uncontrolled arrhythmia requiring pharmacologic therapy;
  4. New York Society of Cardiology classification ≥ grade III; 2. cardiac ejection fraction (LVEF) less than 50%; 3. history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, history of clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormality within 6 months prior to recruitment.
* 4. active hepatitis B or C infection (hepatitis B virus surface antigen positive and hepatitis B virus DNA greater than 1x103 copies/mL; hepatitis C virus RNA greater than 1x103 copies/mL);
* 5. Human Immunodeficiency Virus (HIV) infection (HIV antibody positive);
* 6. imaging confirmation of intestinal obstruction;
* 7. previous or current concurrent other malignancies (except effectively controlled non-melanoma basal cell carcinoma of the skin, carcinoma in situ of the breast/cervix, and other malignancies that have been effectively controlled without treatment within the past five years);
* 8. pregnant and lactating women and patients of childbearing age who do not wish to use contraception;
* 9. patients with other malignant tumors requiring treatment;
* 10. history of pulmonary hemorrhage/coughing up ≥ grade 2 (defined as at least 2.5 mL of bright red blood) within 1 month prior to the first dose;
* 11. a history of arterial embolism, severe hemorrhage (other than hemorrhage due to surgery), or a predisposition to existing embolism or severe hemorrhage within 6 months prior to the first administration of the drug
* 12. a combination of symptomatic brain metastases, meningeal metastases, spinal cord tumor invasion, and spinal cord compression
* 13. use of strong inhibitors or inducers of CYP3A4, CYP2C8, and UGT1A1 within 14 days prior to receiving study drug therapy
* 14. who have used other clinical trial medications within 1 month prior to the first dose;
* 15. female patients who are pregnant or lactating, and subjects of childbearing age who refuse to accept contraceptive measures
* 16. patients who are not suitable for participation in this study in the judgment of the investigator, .-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
(PFS) | 1 year
  Progression-free survival: Defined as time from the date of randomization to first documented disease progression using RECIST version 1.1 by investigator review or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
(ORR) | 1 year
  Objective remission rate:Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1
(DCR) | 1 year
  Disease Control Rate:Defined as the percentage of patients who achieved CR, PR, and stable disease (SD) according to RECIST v1.1
(OS) | 1 year
  Defined as the time between the date of randomization and death due to various causes
Incidence of adverse events | 1 year
  Use NCI-CTCAE version 5.0 for classification and grading

IPD SHARING:
Plan to Share IPD: No